CLINICAL TRIAL: NCT04703283
Title: Effect of a Self-help Smartphone-based Lifestyle Intervention in Reducing Insomnia Symptoms: A Randomized Controlled Trial
Brief Title: Self-help Lifestyle Medicine for Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY012
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Insomnia
Keywords: Insomnia; Lifestyle Medicine; Self-help
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Medicine Group (Experimental): Lifestyle intervention with components including exercise, diet, stress management, and sleep management
  Interventions: Behavioral: Lifestyle Medicine
- Waitlist Control Group (No Intervention): Participants in the waitlist control group will receive the intervention after the immediate post-treatment assessment

INTERVENTIONS:
Behavioral: Lifestyle Medicine — Lifestyle intervention with components including exercise, diet, stress management, and sleep management
  Arms: Lifestyle Medicine Group

SUMMARY:
This study will examine the effects of a self-help smartphone-based multi-component lifestyle medicine intervention (LM) for alleviating insomnia symptoms in a Chinese population. Since a range of lifestyle factors are related to the pathogenesis and progression of insomnia, modifying different lifestyle factors simultaneously, such as diet, exercise, stress, and sleep which are empirically supported by previous reviews, may be effective to reduce insomnia symptoms (Reid et al., 2010; Vedaa et al., 2016). Traditional Chinese nutritional values will be integrated into the smartphone application to increase the acceptability towards the intervention. A prevalence study suggested that self-help interventions are preferred due to the potential stigmatization related to mental health interventions and the high cost of mental health services in Hong Kong (Lee, Tsang, & Kwok, 2007). Nonetheless, to date, only limited self-help interventions that target lifestyle medicine for sleep-related problems are available. Through this study, we aimed to promote evidence-based patient care and improve help-seeking behaviors and access to evidence-based lifestyle interventions for insomnia.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial on the effects of a self-help smartphone-based multi-component lifestyle medicine intervention for reducing insomnia symptoms in the Chinese population. Prior to all study procedures, eligible participants will be required to complete an online informed consent (with telephone support). Assuming an alpha error of 5%, a beta error rate of 20%, and a between-group effect size of 0.77 for the Insomnia Severity Scale (Ip et al., 2020), the final sample is 28 for both groups. With an estimation of 20% withdrawal, 70 eligible participants will be randomly assigned to either the smartphone-based multi-component lifestyle medicine intervention (LM group) or the waitlist control group (WL group) in a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents
* Aged ≥ 18 years
* Have an Insomnia Severity Index (ISI) score ≥10, indicating at least sub threshold level of insomnia symptoms are present
* Able to read Chinese and type in Chinese or English
* Have an Internet-enabled mobile device (iOS or Android operating system)
* Are willing to provide informed consent and comply with the trial protocol

Exclusion Criteria:

* Current involvement in psychotherapy or unstable medication for sleep, depression, and/or anxiety
* Beck Depression Inventory (BDI-II) Item 9 score of at least 2 indicating a current moderate suicidal risk that requires active crisis management (referral information to professional services will be provided to those with serious suicidal risk)
* Are having unsafe conditions and are not recommended for exercise or a change in diet by physicians
* Having major psychiatric, medical, or neurocognitive disorders that make participation infeasible or interfere with the adherence to the lifestyle modification
* Other untreated sleep disorders, including narcolepsy, obstructive sleep apnoea (OSA), and restless leg syndrome (RLS)/periodic leg movement disorder (PLMD) based on the cut-off scores (≥ 7 on narcolepsy; ≥ 15 on OSA; ≥ 7 on RLS/PLMD) of individual sections in SLEEP-50
* Shift work, pregnancy, work, family, or other commitments that interfere with regular night-time sleep patterns
* Hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Change in the Insomnia Severity Index (ISI) | Baseline, immediately post-intervention, and 1-month post-intervention
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.

SECONDARY OUTCOMES:
Change in the Hospital Anxiety and Depression Scale (HADS) | Baseline, immediately post-intervention, and 1-month post-intervention
  The HADS, a self-reporting questionnaire used for assessing the level of depressive and anxiety symptoms over the past week on a 4-point scale. The HADS consists of two parts: an anxiety subscale (HADS-A) and a depression subscale (HADS-D), both of which have seven items.
Change in the Short Form (Six-Dimension) Health Survey (SF-6D) | Baseline, immediately post-intervention, and 1-month post-intervention
  SF-6D is a preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality.
Change in the Health-Promoting Lifestyle Profile (HPLP II) | Baseline, immediately post-intervention, and 1-month post-intervention
  The 52-item HPLPII is composed of a total scale and six subscales to measure behaviors in the theorized dimensions of health-promoting lifestyle: spiritual growth, interpersonal relations, nutrition, physical activity, health responsibility, and stress management.
Change in the Sheehan Disability Scale (SDS) | Baseline, immediately post-intervention, and 1-month post-intervention
  SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life.
Change in the Credibility-Expectancy Questionnaire (CEQ) | Baseline, immediately post-intervention, and 1-month post-intervention
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success.
Change in the Pittsburgh sleep quality index (PSQI) | Baseline, immediately post-intervention, and 1-month post-intervention
  Participants' subjective sleep disturbance over the past month will be assessed using PSQI. PSQI consists of 19 self-rating items that can be categorized into seven components, including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is scored on a 4-point Likert scale (0-3). The sum of the seven components results in a global score of 21. A high score indicates worse sleep quality.
Change in the Consensus Sleep Diary (CSD-M) | Baseline, immediately post-intervention, and 1-month post-intervention
  The standardized sleep diary records sleep time, wake time, perceived sleeping quality, use of hypnotics, etc. on a daily basis. Variables derived from the sleep diary include sleep onset latency (SOL), wake after sleep onset (WASO), total wake time (TWT), total sleep time (TST), sleep efficiency (SE), etc.
Self-developed survey | Baseline
  The self-developed survey will collect information including demographic information (e.g., age, gender, level of education, working industry, relationship status, and location of residence), substance use, body mass index (BMI), rest-activity pattern, and social rhythms, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong